CLINICAL TRIAL: NCT06811883
Title: Optimising Hip Mobility, Hamstring Flexibility and Performance in Elite Sprint and Hurdles Athletes Using Lightback: an Experimental Pilot Study
Brief Title: Optimising Hip Mobility, Hamstring Flexibility and Performance Using Lightback
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica de Ávila (Other)
Responsible Party: Principal Investigator, JORGE VELAZQUEZ SAORNIL, PhD., Universidad Católica de Ávila
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 31/01/2025
Record Dates: First submitted 2025-01-31; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-01

CONDITIONS: Injury;Sports
Keywords: range of motion; prevention; Physiotherapy; athletics
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: LIGHTBACK Group
Who Masked: Participant
Masking Description: Placebo Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LIGHTBACK Gropu (Experimental): This group will perform a standard 20-minute warm-up, and in addition to their usual warm-up, the LIGHTBACK protocol is included.
  Interventions: Device: LIGHTBACK
- Placebo Group (Placebo Comparator): This group will perform a standard 20-minute warm-up, but the LIGHTBACK protocol is not included and a similar placebo is used.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: LIGHTBACK — This group will perform a standard 20-minute warm-up, and the LIGHTBACK protocol is also included.
  Arms: LIGHTBACK Gropu
Device: Placebo — This group will perform a standard 20-minute warm-up, but the LIGHTBACK protocol is not included and a similar placebo is used.
  Arms: Placebo Group

SUMMARY:
In athletics, in the sprint and hurdles disciplines, muscle injuries account for a significant proportion of injuries. The hamstrings are particularly vulnerable, accounting for between 12% and 26% of all injuries in these sports. A single-blind study was conducted on 20 hurdler patients with the intention of assessing hip mobility, hamstring flexibility and performance. To collect this data, the research team will conduct examinations and interviews with the athletes in two groups: an experimental group using LightBack and a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Sprinters and hurdlers aged 18 to 30 years.
* No history of recent (less than 6 months) hamstring or hip injury.
* Signed informed consent.

Exclusion Criteria:

* Cruciate or hamstring tears less than 6 months old;
* Hip and back surgery less than 3 months old;
* Chronic or acute back problems;
* Pregnancy;
* Osteoporosis
* Tumours, bone cancer of the hip and pelvis;
* Direct trauma to the back of the thigh less than 6 months old.
* Orthopaedic or neurological pathologies affecting mobility or muscle activation.
* Participation in another specific training protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
hip mobility | 5 weeks
  measurement of hip mobility measured by goniometry

SECONDARY OUTCOMES:
hamstring flexibility | 5 weeks
  hamstring flexibility measured with inclinometer, in degrees
performance | 5 weeks
  It is a numerical result achieved within the jumping tests: contamovement jump (CMJ): It shall be measured using a force platform with an HD system, which ensures accurate data collection. 0 minimum, 100 maximum.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Pontificia de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Edouard P, Branco P, Alonso JM. Muscle injury is the principal injury type and hamstring muscle injury is the first injury diagnosis during top-level international athletics championships between 2007 and 2015. Br J Sports Med. 2016 May;50(10):619-30. doi: 10.1136/bjsports-2015-095559. Epub 2016 Feb 17. PMID 26887415
- [Result] Askling CM, Tengvar M, Thorstensson A. Acute hamstring injuries in Swedish elite football: a prospective randomised controlled clinical trial comparing two rehabilitation protocols. Br J Sports Med. 2013 Oct;47(15):953-9. doi: 10.1136/bjsports-2013-092165. Epub 2013 Mar 27. PMID 23536466
- [Result] Edouard P, Lahti J, Fleres L, Ahtiainen J, Ulvila JJ, Lehtinen T, Virtanen N, Taipale T, Bellver M, Peltonen V, Thibault M, Huuhka T, Toivonen RM, Morin JB, Mendiguchia J. A musculoskeletal multifactorial individualised programme for hamstring muscle injury risk reduction in professional football: results of a prospective cohort study. BMJ Open Sport Exerc Med. 2024 Feb 8;10(1):e001866. doi: 10.1136/bmjsem-2023-001866. eCollection 2024. PMID 38347859
- [Result] Edouard P, Mendiguchia J, Lahti J, Arnal PJ, Gimenez P, Jimenez-Reyes P, Brughelli M, Samozino P, Morin JB. Sprint Acceleration Mechanics in Fatigue Conditions: Compensatory Role of Gluteal Muscles in Horizontal Force Production and Potential Protection of Hamstring Muscles. Front Physiol. 2018 Nov 30;9:1706. doi: 10.3389/fphys.2018.01706. eCollection 2018. PMID 30555346
- [Result] Bissas A, Paradisis GP, Hanley B, Merlino S, Walker J. Kinematic and Temporal Differences Between World-Class Men's and Women's Hurdling Techniques. Front Sports Act Living. 2022 Apr 29;4:873547. doi: 10.3389/fspor.2022.873547. eCollection 2022. PMID 35571744
- [Result] Nagahara R, Wakamiya M, Shinohara Y, Nagano A. Ground reaction forces during sprint hurdles. J Sports Sci. 2021 Dec;39(23):2706-2715. doi: 10.1080/02640414.2021.1954325. Epub 2021 Jul 27. PMID 34313537